CLINICAL TRIAL: NCT01565720
Title: A Phase 1, Randomized, Double Blind, Placebo and Active Controlled, Parallel Study to Evaluate the Effect of Repeat Doses of Isavuconazole on Cardiac Repolarization in Healthy Adult Subjects
Brief Title: Study of the Effect of Repeat Doses of Isavuconazole on Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 9766-CL-0017
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Pharmacokinetics of Isavuconazole; Healthy Volunteers
Keywords: Isavuconazole; Healthy Volunteers; BAL8557
MeSH Terms: interventions — isavuconazole; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Isavuconazole low dose 3 times per day (TID) for 2 days followed by isavuconazole low dose once a day (QD) for 11 days
  Interventions: Drug: Isavuconazole
- Group 2 (Experimental): Isavuconazole low dose 3 times per day (TID) for 2 days followed by isavuconazole high dose once a day (QD) for 11 days
  Interventions: Drug: Isavuconazole
- Group 3 (Placebo Comparator): Placebo 3 times a day (TID) for 2 days followed by placebo once a day (QD) for 11 days
  Interventions: Drug: Placebo
- Group 4 (Active Comparator): Placebo 3 times a day (TID) for 2 days followed by placebo once a day (QD) for 10 days and then moxifloxacin on Day 13
  Interventions: Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL8557
  Arms: Group 1; Group 2
Drug: Placebo — oral
  Arms: Group 3; Group 4
Drug: Moxifloxacin — oral
  Arms: Group 4

SUMMARY:
This study is designed to evaluate repeat doses of isavuconazole on cardiac repolarization in healthy adult subjects. Eligible subjects will be randomized to one of four treatment groups and be confined for 17 days including pre-dosing days. Moxifloxacin will be given as an active control on the last dosing day to healthy subjects in one of the four groups. All treatments, except the moxifloxacin dose, are double-blinded (neither the subject nor the study doctor will know the treatment assignment). Subjects will undergo continuous ECGs on three study days. ECGs, vital signs, blood draws will be obtained throughout the study for safety and to assess the amount of study drug in body.

ELIGIBILITY:
Inclusion Criteria:

* Subject must weigh at least 45 kg and have a body mass index of 18-30 kg/m2
* If female, the subject agrees to sexual abstinence, is surgically sterile, postmenopausal or using a medically acceptable double-barrier method to prevent pregnancy and agrees to continue using this method during the study and until two weeks after the end of the study. Female subjects must not be lactating or pregnant as documented by a negative pregnancy test at Screening and Day -3
* If male, the subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method during the study and until two weeks after the end of the study
* The subject's clinical laboratory test results at Screening and Day -3 are within normal limits or any abnormal results are considered not to be clinically significant
* The subject has a sitting systolic blood pressure between 90 and 140 mmHg, inclusive and diastolic blood pressure between 50 and 90 mmHg, inclusive at Screening and Day -3
* The subject has good venous access

Exclusion Criteria:

* The subject has a previous history of any clinically significant gastro-intestinal, neurological, renal, hepatic, pulmonary, metabolic, cardio-vascular, psychiatric, endocrine, hematological disorder or disease, malignancy excluding non-melanoma skin cancer or any other medical condition that would preclude participation in the study
* The subject has evidence of any cardiac conduction abnormalities
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia, torsade de pointes, structural heart disease, or family history of Long QT syndrome or Short QT syndrome
* The subject has potassium, calcium, or magnesium levels that are below the clinical laboratory's lower limit of normal
* The subject has a history of consuming more than 14 units of alcoholic beverages per week, has a history of alcohol abuse within the past 2 years prior to Screening, or has a positive screen for alcohol at Screening or Day 3. (NOTE: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor.)
* The subject has a history of drug, chemical, or substance abuse within the past 2 years prior to Screening or has a positive test at Screening or Day -3 for drugs of abuse
* The subject has used tobacco-containing products or nicotine-containing products within 3 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Screening, or over-the-counter medication within 7 days prior to Screening (with the exception of acetaminophen up to 2 grams/day)
* The subject anticipates an inability to abstain from caffeine or alcohol for 48 hours prior to Day -3 and throughout the duration of the study
* The subject anticipates an inability to abstain from grapefruit, Seville oranges, star fruit, or any products containing these items from 72 hours prior to Day -3 and throughout the duration of the study
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 7 days prior to Day -3
* The subject has been vaccinated within the last 30 days prior to Screening
* The subject has a positive test for hepatitis C antibody or hepatitis B surface antigen at Screening or a known history of human immunodeficiency virus
* The subject has known or suspected hypersensitivity to any of the quinolone antibiotics or a history of tendonitis and/or liver function abnormality related to quinolone antibiotic treatment
* The subject has a known or suspected hypersensitivity to isavuconazole, the azole class of compounds, or any components of the study drugs
* The subject has received an experimental agent within 30 days or five half-lives, whichever is longer, prior to Screening
* The subject has had any significant blood loss, donated one or more units (450 mL) of blood or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to Day -3
* The subject has any other condition, which in the opinion of the investigator, precludes the subject's participation in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QT interval corrected for heart rate using Fridericia's correction (QTcF) | Baseline and Day 13

SECONDARY OUTCOMES:
Change from baseline in Electrocardiogram (ECG) variables: QT, PR, RR intervals, QRS, and Heart Rate | Baseline and Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel, Glendale, California, United States